CLINICAL TRIAL: NCT00500123
Title: The Alpha-1 Foundation's and University of Florida's Alpha-1 Coded Testing (ACT) Study
Acronym: ACT
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201903430
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Alpha-1 Antitrypsin Deficiency
Keywords: alpha-1; antitrypsin; AAT; genetic testing; alpha-1 antitrypsin deficiency; AATD
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — A blood card is mailed to the participants home. The provide lancet is used for fingerstick collection of sufficient bloodspots to genotype for alpha-1 antitrypsin (AAT) deficiency alleles and to estimate an AAT level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Alpha-1 Antitrypsin Genotype — Home fingerstick testing for alpha-1 antitrypsin genotype

SUMMARY:
The Alpha-1 Coded Testing (ACT) Study was established to study genetic testing and outcomes of individuals at risk for alpha-1 antitrypsin deficiency.

DETAILED DESCRIPTION:
Genetic testing for alpha-1 antitrypsin deficiency is sometimes delayed despite established testing indications. All genetic tests have risks and possible benefits. The ACT study evaluates the population demographics, reasons for testing, and outcomes through a confidential testing program. Co-morbidities of alpha-1 antitrypsin deficiency other than lung and liver disease are being investigated. Concerns about genetic confidentiality are lessened in this study by a coded testing procedure that returns results through the mail to study participants.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of any age at risk for alpha-1 antitrypsin deficiency on the basis of symptoms or family genetic risk.

Exclusion Criteria:

* Any person who has already had genotype and AAT level testing completed and has a qualified result.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals choosing to test at home for alpha-1 antitrypsin deficiency.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2001-01 (Actual); Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Structured questionnaire responses on the risks and benefits of testing. | Before and after alpha-1 antitrypsin testing
  Rotating questionnaires assess the clinical course and co-morbidities associated with different genotypes of alpha-1 antitrypsin deficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Karina Serban, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coors ME, Moseley R, McGorray S. Informed consent process in Alpha-1 testing of at-risk children: views of parents and adults tested as children. COPD. 2011 Feb;8(1):30-8. doi: 10.3109/15412555.2010.541958. PMID 21299476
- [Background] Holm KE, Borson S, Sandhaus RA, Ford DW, Strange C, Bowler RP, Make BJ, Wamboldt FS. Differences in adjustment between individuals with alpha-1 antitrypsin deficiency (AATD)-associated COPD and non-AATD COPD. COPD. 2013 Apr;10(2):226-34. doi: 10.3109/15412555.2012.719049. PMID 23547634
- [Background] Stoller JK, Strange C, Schwarz L, Kallstrom TJ, Chatburn RL. Detection of alpha-1 antitrypsin deficiency by respiratory therapists: experience with an educational program. Respir Care. 2014 May;59(5):667-72. doi: 10.4187/respcare.02817. Epub 2013 Oct 8. PMID 24106322
- [Result] Strange C, Dickson R, Carter C, Carpenter MJ, Holladay B, Lundquist R, Brantly ML. Genetic testing for alpha1-antitrypsin deficiency. Genet Med. 2004 Jul-Aug;6(4):204-10. doi: 10.1097/01.gim.0000132669.09819.79. PMID 15266208
- [Result] Strange C, Moseley MA, Jones Y, Schwarz L, Xie L, Brantly ML. Genetic testing of minors for alpha1-antitrypsin deficiency. Arch Pediatr Adolesc Med. 2006 May;160(5):531-4. doi: 10.1001/archpedi.160.5.531. PMID 16651497
- [Result] Carpenter MJ, Strange C, Jones Y, Dickson MR, Carter C, Moseley MA, Gilbert GE. Does genetic testing result in behavioral health change? Changes in smoking behavior following testing for alpha-1 antitrypsin deficiency. Ann Behav Med. 2007 Feb;33(1):22-8. doi: 10.1207/s15324796abm3301_3. PMID 17291167
- [Result] McGee D, Strange C, McClure R, Schwarz L, Erven M. The Alpha-1 Association Genetic Counseling Program: an innovative approach to service. J Genet Couns. 2011 Aug;20(4):330-6. doi: 10.1007/s10897-011-9355-z. Epub 2011 Mar 19. PMID 21424325
- See also: Alpha-1 Coded Testing Link — http://www.alphaoneregistry.org